CLINICAL TRIAL: NCT04708977
Title: Is Indirect Decompression Sufficient for the Treatment of Central Stenosis?: A Randomized Controlled Trial
Brief Title: Indirect vs. Direct Decompression for Treatment of Central Stenosis: RCT
Acronym: IDVD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The patient population is too low to conduct the study in a feasible and meaningful amount of time.
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-2228
Record Dates: First submitted 2020-12-22; First posted 2021-01-14 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Patients With Spinal Stenosis Indicated for LLIF
Keywords: Lateral Lumbar Interbody Fusion (LLIF); Foraminal Stenosis; Spine Fusion; Decompression; Lumbar

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized controlled trial.
Who Masked: Participant
Masking Description: Patients will be blinded to randomization and surgical technique will not be evident based on postoperative radiographs. Research coordinators, surgeons, principal investigator (assisting with randomization) and other co-investigators will not be blinded to the type of surgical procedure performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Indirect Decompression (Active Comparator): Lateral lumbar interbody fusion (LLIF), with indirect decompression
  Interventions: Procedure: One-level lateral lumbar interbody fusion with Indirect Decompression
- Group 2: Direct Decompression (Active Comparator): Lateral lumbar interbody fusion (LLIF), with direct decompression
  Interventions: Procedure: One-level lateral lumbar interbody fusion with Direct Decompression

INTERVENTIONS:
Procedure: One-level lateral lumbar interbody fusion with Indirect Decompression — One-level lateral lumbar interbody fusion, with or without percutaneous posterior instrumentation. Thorough discectomy will be performed using lateral access. Fusion will then be performed using lateral access interbody cage and allograft bone graft with or without use of recombinant human bone morphogenic protein 2.
  Arms: Group 1: Indirect Decompression
Procedure: One-level lateral lumbar interbody fusion with Direct Decompression — One-level lateral lumbar interbody fusion, with or without percutaneous posterior instrumentation. Thorough discectomy will be performed using lateral access instruments. Fusion will then be performed using lateral access interbody cage and allograft bone graft with or without use of recombinant human bone morphogenic protein 2.
  Additionally, direct decompression through midline or parasagittal approach will be utilized. A unilateral laminotomy or complete bilateral laminectomy may be performed.
  Arms: Group 2: Direct Decompression

SUMMARY:
This is a prospective, randomized clinical trial of patients undergoing 1-level lateral lumbar spinal fusion. This study seeks to randomize patients indicated for Lateral Lumbar Interbody Fusion (LLIF) into one of two groups: direct decompression and indirect decompression.

DETAILED DESCRIPTION:
While indirect decompression has been largely accepted as a strategy to treat foraminal stenosis, there is some disagreement regarding its efficacy in treating patients with central and lateral recess stenosis. The current study seeks to randomize patients indicated for Lateral Lumbar Interbody Fusion (LLIF) into one of two groups: direct decompression and indirect decompression. Enrolled participants will be evaluated before surgery, during their hospital course and post-operatively at 6 weeks, 3 months, 6 months, 1 and 2 years. Operative details, complications, reoperation rates, patient reported outcomes, clinical and radiographic outcome measures will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Fusion indicated by the treating surgeon. Fusion may be indicated for one or more of the following reasons:

  * Mobile degenerative spondylolisthesis
  * Severe vertical foraminal stenosis
  * Adjacent segment degeneration and/or degenerative disc disease with suspected discogenic pain
* One-level central canal stenosis

  * WITH neurogenic claudication
  * As measured in preoperative MRI
* Oswestry Low Back Pain Disability Questionnaire score > 35% (18/50)
* Failed 3 months of conservative treatment
* Willing to give written informed consent and psychosocially, mentally, and physically able to comply fully with protocol, including adhering to follow-up schedule and requirements, and filling out forms

Exclusion Criteria:

* Multilevel central canal stenosis
* Patients with vertebral endplate dimensions that are too small to allow for safe placement of an intervertebral cage
* Known allergy to titanium, polyethylene, cobalt, chromium, or molybdenum
* Prior surgery at index disc level (discectomy, decompression, or fusion)
* History of spinal or vertebral infection of the lumbar spine
* History of vertebral fracture of the lumbar spine
* Current pregnancy or interest in becoming pregnant over the next 1 year
* Active infection-systemic or local
* Non-English speakers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Up to 12 months post-operatively
  Change in Oswestry Disability Index (ODI) 100 point scale. The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools [1].
  For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. If all 10 sections are completed the score is calculated by adding all scores for each statement, divided by 50 total possible points, and then multiplied by 100 for a percentage. Percentage scores are interpreted on a scale from 0-20% as minimal disability to 61-100% as crippled.
Comparison of Oswestry Disability Index (ODI) | Up to 24 months post-operatively. (6 weeks, 3, 6, 12, and 24 months timepoints)
  Compare ODI scores to assess the kinetics of improvement in the control (direct decompression) vs. treatment (indirect decompression) groups.
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools [1].
  For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. If all 10 sections are completed the score is calculated by adding all scores for each statement, divided by 50 total possible points, and then multiplied by 100 for a percentage. Percentage scores are interpreted on a scale from 0-20% as minimal disability to 61-100% as crippled.

SECONDARY OUTCOMES:
Reoperation Rate | Within 12 months and 24 months, post-operatively.
  Reoperation rate on the lumbar spine within 12 months and within 24 months
Complication Rate | Within 12 months and 24 months, post-operatively.
  Complication rate within 12 months and within 24 months
Numeric Rated Scale (NRS)-Back and Leg pain | 6- Weeks, 3-, 6-, 12-, and 24-Months.
  Patient Reported Outcomes: Numeric Rated Scale (NRS)-back and leg pain scores
Radiographic Measurements - Lumbar Lordosis | Preoperative and 12-Month radiographs
  Radiographic measurements at 12 months will be compared to preoperative measurements to quantify the change in lumbar lordosis as a result of Lateral Lumbar Interbody Fusion (LLIF). Measurements will be taken in millimeters by (2) co-investigators.
Radiographic Measurements - Segmental Lordosis | Preoperative and 12-Month radiographs
  Radiographic measurements at 12 months will be compared to preoperative measurements to quantify the change in segmental lordosis as a result of Lateral Lumbar Interbody Fusion (LLIF). Measurements will be taken in millimeters by (2) co-investigators.
Radiographic Measurements - Disc Space Height | Preoperative and 12-Month radiographs
  Radiographic measurements at 12 months will be compared to preoperative measurements to quantify the change in disc space height as a result of Lateral Lumbar Interbody Fusion (LLIF). Measurements will be taken in millimeters by (2) co-investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Sravisht Iyer, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only the PI, study coordinators listed on the IRB protocol, and co-investigators will have access to the IPD information.

REFERENCES:
- [Background] Grant S, Aitchison T, Henderson E, Christie J, Zare S, McMurray J, Dargie H. A comparison of the reproducibility and the sensitivity to change of visual analogue scales, Borg scales, and Likert scales in normal subjects during submaximal exercise. Chest. 1999 Nov;116(5):1208-17. doi: 10.1378/chest.116.5.1208. PMID 10559077
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Fujibayashi S, Hynes RA, Otsuki B, Kimura H, Takemoto M, Matsuda S. Effect of indirect neural decompression through oblique lateral interbody fusion for degenerative lumbar disease. Spine (Phila Pa 1976). 2015 Feb 1;40(3):E175-82. doi: 10.1097/BRS.0000000000000703. PMID 25394317
- [Background] Isaacs RE, Sembrano JN, Tohmeh AG; SOLAS Degenerative Study Group. Two-Year Comparative Outcomes of MIS Lateral and MIS Transforaminal Interbody Fusion in the Treatment of Degenerative Spondylolisthesis: Part II: Radiographic Findings. Spine (Phila Pa 1976). 2016 Apr;41 Suppl 8:S133-44. doi: 10.1097/BRS.0000000000001472. PMID 26839992
- [Background] Kono Y, Gen H, Sakuma Y, Koshika Y. Comparison of Clinical and Radiologic Results of Mini-Open Transforaminal Lumbar Interbody Fusion and Extreme Lateral Interbody Fusion Indirect Decompression for Degenerative Lumbar Spondylolisthesis. Asian Spine J. 2018 Apr;12(2):356-364. doi: 10.4184/asj.2018.12.2.356. Epub 2018 Apr 16. PMID 29713419
- [Background] Nakashima H, Kanemura T, Satake K, Ishikawa Y, Ouchida J, Segi N, Yamaguchi H, Imagama S. Indirect Decompression on MRI Chronologically Progresses After Immediate Postlateral Lumbar Interbody Fusion: The Results From a Minimum of 2 Years Follow-Up. Spine (Phila Pa 1976). 2019 Dec 15;44(24):E1411-E1418. doi: 10.1097/BRS.0000000000003180. PMID 31365515
- [Background] Pimenta L. Less-invasive lateral lumbar interbody fusion (XLIF) surgical technique: video lecture. Eur Spine J. 2015 Apr;24 Suppl 3:441-2. doi: 10.1007/s00586-015-3948-4. No abstract available. PMID 25904416
- [Background] Ozgur BM, Aryan HE, Pimenta L, Taylor WR. Extreme Lateral Interbody Fusion (XLIF): a novel surgical technique for anterior lumbar interbody fusion. Spine J. 2006 Jul-Aug;6(4):435-43. doi: 10.1016/j.spinee.2005.08.012. PMID 16825052
- [Background] Smith ZA, Sugimoto K, Lawton CD, Fessler RG. Incidence of lumbar spine pedicle breach after percutaneous screw fixation: a radiographic evaluation of 601 screws in 151 patients. J Spinal Disord Tech. 2014 Oct;27(7):358-63. doi: 10.1097/BSD.0b013e31826226cb. PMID 22688617
- [Background] Baird EO, McAnany SJ, Overley S, Skovrlj B, Guzman JZ, Qureshi SA. Accuracy of Percutaneous Pedicle Screw Placement: Does Training Level Matter? Clin Spine Surg. 2017 Jul;30(6):E748-E753. doi: 10.1097/BSD.0000000000000274. PMID 28632564
- [Background] Sellin JN, Mayer RR, Hoffman M, Ropper AE. Simultaneous lateral interbody fusion and pedicle screws (SLIPS) with CT-guided navigation. Clin Neurol Neurosurg. 2018 Dec;175:91-97. doi: 10.1016/j.clineuro.2018.10.013. Epub 2018 Oct 23. PMID 30384122
- [Background] Houten JK, Nasser R, Baxi N. Clinical assessment of percutaneous lumbar pedicle screw placement using theO-arm multidimensional surgical imaging system. Neurosurgery. 2012 Apr;70(4):990-5. doi: 10.1227/NEU.0b013e318237a829. PMID 21946509
- [Background] Jain D, Manning J, Lord E, Protopsaltis T, Kim Y, Buckland AJ, Bendo J, Fischer C, Goldstein J. Initial Single-Institution Experience With a Novel Robotic-Navigation System for Thoracolumbar Pedicle Screw and Pelvic Screw Placement With 643 Screws. Int J Spine Surg. 2019 Oct 31;13(5):459-463. doi: 10.14444/6060. eCollection 2019 Oct. PMID 31741833
- [Background] Huntsman KT, Riggleman JR, Ahrendtsen LA, Ledonio CG. Navigated robot-guided pedicle screws placed successfully in single-position lateral lumbar interbody fusion. J Robot Surg. 2020 Aug;14(4):643-647. doi: 10.1007/s11701-019-01034-w. Epub 2019 Oct 17. PMID 31625074
- [Background] Boukebir MA, Berlin CD, Navarro-Ramirez R, Heiland T, Scholler K, Rawanduzy C, Kirnaz S, Jada A, Hartl R. Ten-Step Minimally Invasive Spine Lumbar Decompression and Dural Repair Through Tubular Retractors. Oper Neurosurg. 2017 Apr 1;13(2):232-245. doi: 10.1227/NEU.0000000000001407. PMID 28927213
- [Result] Sembrano JN, Tohmeh A, Isaacs R; SOLAS Degenerative Study Group. Two-year Comparative Outcomes of MIS Lateral and MIS Transforaminal Interbody Fusion in the Treatment of Degenerative Spondylolisthesis: Part I: Clinical Findings. Spine (Phila Pa 1976). 2016 Apr;41 Suppl 8:S123-32. doi: 10.1097/BRS.0000000000001471. PMID 26825788
- [Result] Hung M, Saltzman CL, Kendall R, Bounsanga J, Voss MW, Lawrence B, Spiker R, Brodke D. What Are the MCIDs for PROMIS, NDI, and ODI Instruments Among Patients With Spinal Conditions? Clin Orthop Relat Res. 2018 Oct;476(10):2027-2036. doi: 10.1097/CORR.0000000000000419. PMID 30179950